CLINICAL TRIAL: NCT00006126
Title: Allogeneic Peripheral Blood Progenitor Cell Transplantation in Patients With Incurable Solid Tumors: A Phase I Study
Brief Title: Peripheral Stem Cell Transplantation in Treating Patients With Melanoma or Small Cell Lung, Breast, Testicular, or Kidney Cancer That is Metastatic or That Cannot Be Treated With Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to accrue subjects.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Richard Burt, MD, Northwestern University
Purpose: Treatment
Other Study IDs: NU 99H2; NU-99H2; NCI-G00-1838
Record Dates: First submitted 2000-08-03; First posted 2004-03-08 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer; Kidney Cancer; Lung Cancer; Melanoma (Skin); Testicular Germ Cell Tumor
Keywords: stage IV breast cancer; recurrent breast cancer; stage IV renal cell cancer; recurrent renal cell cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage II malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Breast Neoplasms; Kidney Neoplasms; Lung Neoplasms; Melanoma; Testicular Germ Cell Tumor; Carcinoma, Renal Cell; Small Cell Lung Carcinoma; Testicular Neoplasms | interventions — Busulfan; Cyclophosphamide; Etoposide; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: etoposide
Drug: fludarabine phosphate
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of peripheral stem cell transplantation in treating patients who have melanoma or small cell lung, breast, testicular, or kidney cancer that is metastatic or that cannot be treated with surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of allogeneic peripheral blood stem cell transplantation in patients with metastatic or unresectable small cell lung cancer, breast cancer, testicular germ cell cancer, melanoma, or renal cell cancer. II. Determine the efficacy of this regimen in these patients.

OUTLINE: Donors receive filgrastim (G-CSF) subcutaneously for 4 or 5 days prior to peripheral blood stem cell harvest. Patients are assigned to one of three conditioning regimens, depending on disease. Group A (small cell lung cancer): Patients receive cyclophosphamide IV over 1-2 hours on days -7 and -6, etoposide IV over 4 hours on day -5, and total body irradiation twice daily on days -4 to -1. Group B (breast cancer and testicular germ cell cancer): Patients receive oral busulfan every 6 hours on days -7 to -4 for a total of 14 doses. Patients then receive cyclophosphamide IV over 1-2 hours on days -3 and -2. Group C (renal cell cancer and melanoma): Patients receive fludarabine IV daily on days -8 to -4 and cyclophosphamide IV on days -3 and -2. All groups: Patients receive allogeneic peripheral blood stem cells IV over 10-20 minutes on day 0. Patients are followed weekly for 3 months, at 6 and 12 months, and then yearly for 5 years.

PROJECTED ACCRUAL: A total of 19-42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic or unresectable solid tumor of one of the following types: Small cell lung cancer Extensive stage (disease outside the hemithorax) or relapsed Prior cytoreduction with platinum/etoposide regimen and/or taxane containing regimen Epithelial breast cancer Stage IV or relapsed disease Prior cytoreduction with adriamycin and/or taxane regimens Testicular germ cell cancer Failure to achieve complete remission with platinum based chemotherapy Relapsed disease with at least one salvage regimen Melanoma Metastatic disease that has failed at least one biologic response modifier such as interleukin-2 or interferon Relapsed disease involving a visceral organ Renal cell cancer Metastatic disease that has failed at least one biologic response modifier such as interleukin-2 or interferon Relapsed disease involving a visceral organ HLA matched or one antigen mismatched related donor available Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Under physiologic 60 Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL unless due to Gilbert's disease SGOT no greater than 3 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No congestive heart failure LVEF at least 40% Pulmonary: DLCO at least 45% of predicted OR FEV1/FVC at least 50% of predicted Other: HIV negative Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy that would preclude study Surgery: See Disease Characteristics

Max Age: 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 1999-09; Primary Completion 2001-04; Study Completion 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Richard K. Burt, MD, Study Chair — Robert H. Lurie Cancer Center